CLINICAL TRIAL: NCT05554432
Title: Development of an EORTC Immune Checkpoint Inhibitor-specific Quality of Life Item List: Phase 1 & 2
Acronym: EORTC ICI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: IC 2022-03
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Cancer; IMMUNE CHECKPOINT INHIBITOR; Quality of Life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Over the past 20 years, the views and experiences of patients in the field of oncology (through patient-reported outcomes, PROMs) have become increasingly important. When used in clinical trials, PROMs contribute to better detection and are used in clinical trials to improve the detection and management of treatment side effects. The Health-related quality of life assessments are widely used in oncology research, and the development of reliable and valid measurement instruments has become a major challenge.

In this context, health-related quality of life in cancer patients covers various aspects (functional status, physical or psychological symptoms) and several cancer-specific measurement instruments have been developed, including the EORTC QLQ-C30 quality of life questionnaire.

Among the different therapies used to treat cancers, immunotherapy with immune checkpoint inhibitors has been gaining momentum in recent years. Commonly used to treat a wide variety of cancers, it also has a wide range of known side effects.

However, little is known about the health-related quality of life of patients patients who receive this therapy: specific self-questionnaires are almost non-existent or inadequate, not covering all the effects related to immune checkpoint inhibitor toxicity. As for the data currently collected, they suffer from methodological problems.

In view of the increasing use of immune checkpoint inhibitors in cancer treatment, their known side effects and the lack of valid questionnaires specific to these treatments, it appears important to provide a valid questionnaire to take into account these impacts on the quality of life of patients.

ELIGIBILITY:
Patients :

Inclusion Criteria:

* Provision of written informed consent to participate in the study
* Has been diagnosed with cancer
* Either currently receiving, or has received in the previous 12 months, one of the following:

  * an anti-PD-1 or anti-PDL-1 agent as the sole immune checkpoint inhibitor treatment (at least three cycles)
  * an anti-PD-1 or anti-PDL-1 agent in combination with an anti-CTLA-4 agent (at least one cycle)
  * cytotoxic chemotherapy and an anti-PD-1 or anti-PDL-1 agent (at least three cycles)
* Aged ≥18 years

Exclusion Criteria:

* Has an additional primary cancer for which they are receiving systemic therapy
* Cognitive impairment which presents an obstacle to the completion of questionnaires or an interview
* Poor command of the locally dominant language, or an inability to read questions
* [Phase 1b only] Was interviewed for Phase 1a

Healthcare professionals :

Inclusion Criteria:

* Holds, or has held, a professional clinical position which involves working directly with cancer patients who are in receipt of immune checkpoint inhibitors
* Is a medical oncologist, nurse specialist (or equivalent), psychologist, or social worker

Exclusion Criteria:

• Has met the inclusion criteria for <1 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patient population is individuals aged over 18, with a diagnosis of cancer, who have received or are receiving treatment with one of the following:
  * anti-PD-1 (e.g., nivolumab, pembrolizumab, cemiplimab) or anti-PDL-1 (e.g., atezolizumab, avelumab, durvalumab) only
  * anti-PD-1 + anti-CTLA-4 (e.g., nivolumab + ipilumumab) only
  * anti-PD-1/anti-PDL-1 + chemotherapy
  Experienced HCPs who have worked with patients who have received or are receiving ICIs will be eligible for inclusion, in line with the EORTC QLG guidelines which state that HCPs should be interviewed for their views on HRQoL issues affecting these patients.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
To assess the need for an additional EORTC quality of life module, or item list, to measure health-related quality of life in cancer patients who have received or are receiving immune checkpoint inhibitors. | At inclusion
  Provisional item list(s) of quality of life issues important to people treated with immune checkpoint inhibitors.
  Development of a strategy for the measurement of health-related quality of life in cancer patients who have received immune checkpoint inhibitors, alongside existing EORTC quality of life scales for cancer patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Curie, Paris, France